CLINICAL TRIAL: NCT06274164
Title: Clinical and Molecular Biomarker Studies in RAI1-Related Disorders
Brief Title: Clinical and Molecular Biomarker Studies in RAI1 (Retinoic Acid-Induced 1) -Related Disorders
Status: Recruiting | Type: Observational
Sponsor: Baylor College of Medicine (Other)
Collaborators: Doris Duke Charitable Foundation (Other)
Responsible Party: Principal Investigator, Davut Pehlivan, MD, Assistant Professor, Pediatrics-Neurology, Baylor College of Medicine
Other Study IDs: H-54820 / RAI1
Record Dates: First submitted 2024-02-16; First posted 2024-02-23 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: RAI1 Gene 17P11.2 Deletion+Duplication
Keywords: Smith-Magenis syndrome (SMS); Potocki-Lupski Syndrome (PTLS); RAI1-related disorders; Retinoic Acid-Induced 1-related disorders
MeSH Terms: conditions — Smith-Magenis Syndrome; Potocki-Lupski syndrome | interventions — Electroencephalography; Polysomnography; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Optional Skin biopsy will performed and used to generate cell lines.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patient group: Subject enrollment: patients with RAI1-related disorders will be enrolled and will complete the following assessments:
  * Clinical studies: vitals, history and physical examinations.
  * Neurophysiological studies: sleep/EEG study (for a selected patient population).
  * Molecular (biomarkers) studies: blood (required) and skin biopsy (optional).
  Interventions: Diagnostic Test: Electroencephalography/Polysomnography (EEG/PSG); Procedure: Skin Biopsy; Diagnostic Test: Blood draw
- Control group: Subject enrollment: healthy family members of the patients with RAI1-related disorders who are willing to give a blood sample.
  Molecular (biomarkers) studies: blood samples will be used as healthy control for biomarker studies.
  Interventions: Diagnostic Test: Blood draw

INTERVENTIONS:
Diagnostic Test: Electroencephalography/Polysomnography (EEG/PSG) — Instigators will determine if subjects are candidate for the procedure. A sleep study records the brain electrical waves, the oxygen level in the blood, heart rate breathing, as well as eye and leg movements. Subjects will need to be admitted overnight for the sleep study.
  Other Names: sleep study
  Groups: Patient group
Procedure: Skin Biopsy — A special 3-4 mm (0.12 inches) wide circular tool will be used to remove a small section of skin including deeper layers. A numbing cream or injectable anesthetic (i.e. lidocaine) will be applied to the area before the procedure. Sample will be used to create a cell line. This means that investigators would treat the cells from the sample in a way that allows to grow them in the laboratory. Investigators will then use these cells in research.
  Groups: Patient group
Diagnostic Test: Blood draw — A single blood sample of 15 cc (not exceeding 3 cc per kg) (~3 teaspoons) will be collected for metabolomics (biomarker) study. From available family members, same amount of blood will be obtained to use as a control sample.

SUMMARY:
Currently, there is no clinically available genetic-based treatment for RAI1 (Retinoic Acid-Induced 1) -related disorders other than symptomatic management and there are no established clinical or molecular biomarkers that could be used as measures for the efficacy of therapy in future treatment studies. Biomarkers are measures of what is happening inside the body, shown by the results of laboratory, imaging or other tests.

Biomarkers can help doctors and scientists diagnose diseases and health conditions, monitor responses to treatment and see how a person's disease or health condition changes over time.

The goal of this observational and laboratory study is to develop clinical, neurophysiology and molecular biomarkers in RAI1-related disorders. The main question[s] it aims to answer are:

* to characterize the disease features more precisely and analyze the differentiating and overlapping features of RAI1-related disorders (Smith-Magenis syndrome and Potocki-Lupski Syndrome)
* to identify clinical, neurophysiology, and laboratory biomarkers that differentiate RAI1-related disorders one from another.

Participants will have to complete:

* a clinical examination
* a blood draw
* a skin biopsy (optional)
* a sleep study

Researchers will compare patients' blood to control group's blood for biomarker studies.

DETAILED DESCRIPTION:
20 SMS (Smith-Magenis syndrome) patients and 20 PTLS (Potocki-Lupski Syndrome) patients will be enrolled in the study. Additionally, up to 50 healthy controls will be enrolled among family members of patients.

All the assessments may be completed during a one-time visit at the hospital which includes an overnight stay for the sleep study for selected individuals. In case all the procedures could not be completed during the one-time visit, subjects may be asked to come again for the remaining procedure.

Tests, procedures and samples to be completed or collected:

* Demographics will be collected
* History and physical examination: A detailed birth, medical, surgical and medication history will be collected as well as seizure and movement disorder histories. Subject chart will be reviewed to complete this data collection. A general physical examination and detailed neurological examination will be performed.
* Vitals: blood pressure, temperature, respiratory rate, weight and height will be collected.
* Polysomnography/electroencephalography (PSG/EEG): clinician Investigator will determine if subject is candidate for the procedure. A sleep study records the brain electrical waves, the oxygen level in the blood, heart rate and breathing, as well as eye and leg movements. Subject will need to be admitted overnight for the sleep study. The exam is video recorded.
* Blood samples: A single blood sample of 15 cc (not exceeding 3 cc per kg) (~3 teaspoons) will be collected for research purposes. Samples will be kept up to 2 years after the study results are published.
* Optional skin biopsy: a skin biopsy from the upper, inner arm, lateral upper thigh, or another area, may be performed for research purposes. A special 3-4 mm (0.12 inches) wide circular tool will be used to remove a small section of skin including deeper layers. A numbing cream or injectable anesthetic (i.e. lidocaine) will be applied to the area before the procedure. Sample will be used to create a cell line. This means that investigators would treat the cells from the sample in a way that allows to grow them in the laboratory. Investigators will then use these cells in research.

ELIGIBILITY:
Inclusion Criteria:

* Patient group:

  * Patients who have RAI1-related disorder confirmed by genetic testing including karyotyping, fluorescence in situ hybridization (FISH), array Comparative Genomic Hybridization (aCGH), single nucleotide polymorphism (SNP) array and next generation sequencing performed by a Clinical Laboratory Improvement Amendments (CLIA)-certified laboratory.
  * Grossly intact hearing and vision as per parent report
  * Age between 1 month to 60 years old
  * Able to complete the study (i.e., travel to site and spend 1 day in Houston)
  * Caregiver with spoken and written English at a level adequate to give informed assent (consent on behalf of the patient) for participation.

Control group:

* Healthy family member, not having a RA1-related disorder
* Age between 5 years to 80 years old

Exclusion Criteria:

* Patient group:

  * Contraindication for blood draw or skin biopsy as determined by the enrolling provider (e.g., bleeding diathesis)
  * Patients who are at high risk including ventilator/tracheostomy dependent, poorly controlled endocrine disorders, and unstable seizures (will be assessed by neurologist), end-stage renal disease.
  * Participation in any investigational treatment study

Control group:

• Patients who have RAI1-related disorder confirmed by genetic testing.

Ages: 1 Month to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with RAI1-related disorders who are willing to participate in clinical, neurophysiological and molecular studies, will be enrolled, as well as healthy family controls. Subjects will have to travel to Texas Children's Hospital to complete study activities.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2024-03-13 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Rate of neurological clinical finding | 2029
  Identify biomarkers which have suitable stability for use in clinical settings by combining quantitative comparisons from the visit with qualitative literature/retrospective chart review synthesis, to prioritize measures for inclusion in a panel of candidate biomarkers.
  Investigators expect to find a clinical exam finding such as tremor which can be measurable objectively or behavior which can be relied on caregiver's report.
Rate of electroencephalogram (EEG) and/or sleep abnormalities | 2029
  Identify biomarkers which have suitable stability for use in clinical settings by combining quantitative comparisons from the visit with qualitative literature/retrospective chart review synthesis, to prioritize measures for inclusion in a panel of candidate biomarkers. To identify candidate oscillatory circuitry biomarkers of Smith-Magenis syndrome (SMS) and Potocki-Lupski Syndrome (PTLS), investigators will use EEG and sleep metrics.
Concentration of downstream molecular pathway interactors of RAI1 | 2029
  Identify biomarkers which have suitable stability for use in clinical settings by combining quantitative comparisons from the visit with qualitative literature synthesis, to prioritize measures for inclusion in a panel of candidate biomarkers.
  There are no biomarkers that trace disease stage and severity in RAI1-related disorders. Towards this goal, investigators aimed to identify molecular biomarkers from patients' plasma by quantifying metabolites.

CONTACTS AND LOCATIONS:
Overall Officials: Davut Pehlivan, MD, Principal Investigator — Texas Children's Hospital - Baylor College of Medicine
Locations (1):
- Texas Children's Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No